CLINICAL TRIAL: NCT05766813
Title: A Randomized, Double-blind, Placebo-controlled Multicenter Study to Assess the Efficacy and Safety of Lenrispodun as Adjunctive Therapy in the Treatment of Patients With Motor Fluctuations Due to Parkinson's Disease
Brief Title: Lenrispodun as Adjunctive Therapy in the Treatment of Patients With Motor Fluctuations Due to Parkinson's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITI-214-202
Record Dates: First submitted 2023-02-24; First posted 2023-03-13 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Parkinson Disease
Keywords: levodopa-induced dyskinesia; ON and OFF state
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lenrispodun 30 mg (Experimental): Lenrispodun 30 mg tablets administered orally, once-daily.
  Interventions: Drug: Lenrispodun
- Placebo (Placebo Comparator): Matching tablets administered orally, once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lenrispodun — Lenrispodun 30 mg tablets administered orally, once daily.
  Arms: Lenrispodun 30 mg
Drug: Placebo — Matching tablets administered orally, once daily.
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group, fixed-dose study in patients with a diagnosis of Parkinson's Disease consistent with the UK Parkinson's Disease Society (UKPDS) Brain Bank diagnostic criteria, who are experiencing wearing off symptoms and levodopa-induced dyskinesia.

DETAILED DESCRIPTION:
The study will be conducted in three periods:

* Screening Period (up to 4 weeks) during which patient eligibility will be assessed;
* Double-blind Treatment Period (4 weeks) in which all patients will be randomized to receive placebo or Lenrispodun 30 mg/day in 1:1 ratio.
* Safety Follow-up Period (1 week) in which all patients will return to the clinic for a safety follow-up visit approximately one week after the last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 40 years of age and older
2. Body mass index of 19.0-40.0 kg/m2;
3. Diagnosis of PD that is consistent with the UK Parkinson's Disease Society (UKPDS) Brain Bank diagnostic criteria;
4. Hoehn and Yahr Scale stage classification of 2 or 3 when in the ON state;
5. Have a clinically meaningful response to levodopa (levodopa + DDCI combination) based on Investigator assessment, and meet the following:

   1. Have been on a stable and optimal dose of levodopa (levodopa + DDCI combination: minimum dose of levodopa equivalent to 100 mg three times daily) for at least 4 weeks prior to Screening, and are expected to continue the same dose regimen throughout the Double-blind Treatment Period;
   2. If taking other anti-parkinsonian medications (MAO-B [monoamine oxidase B] inhibitor, COMT [catechol-O-methyltransferase] inhibitor, dopamine agonist) in addition to levodopa, have been on a stable dose for at least 4 weeks prior to Screening and are expected to continue the same dose regimen throughout the Double-blind Treatment Period;

7. Have wearing-off symptoms and levodopa-induced dyskinesia as per Investigator judgment; 8. Properly complete and return a self-reported home diary for motor function status (Hauser Diary) during the Screening Period, which confirms 3 days (ie, 3 consecutive, 24-hour periods) immediately prior to Baseline, each with at least 2½ hours of OFF time during waking hours.

9. Has a caregiver to assist with study participation, if determined by the Investigator to be necessary.

Exclusion Criteria:

1. Medical history indicating parkinsonism other than idiopathic PD, including but not limited to, progressive supranuclear gaze palsy, multiple system atrophy, drug-induced parkinsonism, essential tremor, primary dystonia;
2. Has late-stage PD, severe peak-dose dyskinesia, clinically significant end-dose or biphasic dyskinesia, and/or unpredictable or widely swinging fluctuations in their symptoms as assessed by the Investigator;
3. Exhibits clinical signs of dementia as indicated by the Mini-Mental State Examination, 2nd Edition: Standard Version (MMSE-2:SV) score of ≤ 24;
4. Use of moderate or strong CYP3A4 inhibitors within 5 half-lives of Baseline or CYP3A4 inducers within 2 weeks of Baseline;
5. Daily use of nonsteroidal anti-inflammatory drugs (NSAIDs), with the exception of acetylsalicylic acid (ASA);
6. Use of MAO-A inhibitors, phosphodiesterase type 5 (PDE5) inhibitors, or alpha blockers including tamsulosin, within 5 half-lives of Baseline;

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Hauser Diary | Day 29
  The Hauser Diary is a validated and commonly used patient-self-report home diary to assess motor symptoms in PD. It asks patients to characterize their predominant motor states in 30-minute intervals as Asleep, OFF, ON without dyskinesia, ON with non-troublesome dyskinesia, and ON with troublesome dyskinesia.

SECONDARY OUTCOMES:
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | Day 29
  The MDS-UPDRS evaluates various aspects of Parkinson's disease and has four parts: Part I (Non-motor Aspects of Experiences of Daily Living), Part II (Motor Aspects of Experiences of Daily Living), Part III (Motor Examination), and Part IV (Motor Complications). The MDS-UPDRS evaluates various aspects of Parkinson's disease and has four parts: Part I (Non-motor Aspects of Experiences of Daily Living), Part II (Motor Aspects of Experiences of Daily Living), Part III (Motor Examination), and Part IV (Motor Complications).
  Each parkinsonian sign or symptom on the MDS-UPDRS is rated on a 5-point scale (ranging from 0 to 4), with higher scores indicating more severe impairment. The maximum total UPDRS score is 199, indicating the worst possible disability from PD.

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Clinical Site, Phoenix, Arizona
  - Clinical Site, Scottsdale, Arizona
  - Clinical Site, Irvine, California
  - Clinical Site, Loma Linda, California
  - Clinical Site, Altamonte Springs, Florida
  - Clinical Site, Boca Raton, Florida
  - Clinical Site, Coral Springs, Florida
  - Clinical Site, Hallandale, Florida
  - Clinical Site, Maitland, Florida
  - Clinical Site, Miami, Florida
  - Clinical Site, Ocala, Florida
  - Clinical Site, Orlando, Florida
  - Clinical Site, Port Orange, Florida
  - Clinical Site, Tampa, Florida
  - Clinical Site, Augusta, Georgia
  - Clinical Site, Decatur, Georgia
  - Clinical Site, Kansas City, Kansas
  - Clinical Site, Farmington Hills, Michigan
  - Clinical Site, Golden Valley, Minnesota
  - Clinical Site, Albany, New York
  - Clinical Site, Rock Hill, South Carolina
  - Clinical Site, Memphis, Tennessee
  - Clinical Site, Austin, Texas
  - Clinical Site, Dallas, Texas
  - Clinical Site, Georgetown, Texas
  - Clinical Site, Falls Church, Virginia
  - Clinical Site, Henrico, Virginia
  - Clinical Site, Kirkland, Washington
  - Clinical Site, Spokane, Washington
  - Clinical Site, Milwaukee, Wisconsin